CLINICAL TRIAL: NCT01528150
Title: Clinical Investigation to Assess the Safety and Efficacy of the Tendril MRI™ Leads, as a Part of the Accent MRI™ System, in Patients With Standard Bradycardia Pacing Indication.
Brief Title: Safety and Efficacy Study of Tendril MRI™ Leads in Standard Bradycardia Pacing Indication
Acronym: TendrilMRI™
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-11-054-EU-LV
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Accent MRI System: Accent MRI system will be implanted = Accent MRI Pacemaker + Tendril MRI Leads

SUMMARY:
The purpose of this observational study is the assessment (safety and efficacy) of the St. Jude Medical Tendril MRI™ leads. The Tendril MRI™ leads are a full part of the Accent MRI™ System, consisting of Tendril MRI™ leads and Accent MRI™ pacemaker. The subject population includes patients with a standard bradycardia pacing indication.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is a diagnostic method to view high quality two and three dimensional images of the body. However, magnetic resonance imaging systems generate three electromagnetic fields that are used to produce an image. These include a static magnetic field, a time varying gradient magnetic field, and a radiofrequency field. All three of these fields interact with implanted devices and could create hazards for the device, the patient, or both. Due to these issues, currently marketed pacemaker systems may be contraindicated for use in an MRI environment.

St. Jude Medical has developed a system, the Accent MRI™ system, comprised of the Accent MRI™ device and the Tendril MRI™ lead, and an investigational MRI Activator™, designed to mitigate such interactions.

ELIGIBILITY:
Inclusion Criteria:

* Approved Class I or Class II indication per: European Society of Cardiology (ESC) guidelines for implantation of a dual chamber pacemaker or single chamber pacemaker, OR American College of Cardiology (ACC) / American Heart Association (AHA) / Heart Rhythm Society (HRS) guidelines for implantation of a dual chamber pacemaker or single chamber pacemaker
* Require a new Accent MRI™ pacemaker and Tendril MRI™ lead (either initial implant or complete system change out with no abandoned devices).
* Is ≥ 18 years of age.
* Able to provide written informed consent prior to any investigational related procedure.
* Willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

* Have an existing pacemaker or ICD (abandoned devices and/or leads are not allowed. A new pacemaker and lead or complete system change out is required for enrollment).
* Have an existing active implanted medical device (e.g., Implantable Cardioverter Defibrillator (ICD), neurostimulator, etc.).
* Have a non-MRI compatible device or material implant (e.g., intracranial aneurysm clip, non-MRI compatible devices or material, metals or alloys, etc.).
* Have a lead extender, plug or adaptor.
* Have a prosthetic tricuspid heart valve.
* Are currently participating in another investigational device or drug investigation.
* Are allergic to Dexamethasone sodium phosphate (DSP).
* Are pregnant or planning to become pregnant during the duration of the study.
* Have a life expectancy of less than 12 months from Screening due to any life-threatening condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: standard bradycardia indications
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob RW Breedveld, MD, Principal Investigator — Medical Center Leeuwarden, the Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Accent MRI System
Started | 466
Completed | 422
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | Accent MRI System
Number analyzed (Participants) | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.74 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 272
AtrioVentricular-Block (AV-Block) [Number; unit: participants]
  No AV Block | 179
  1st Degree AV Block | 41
  2nd Degree AV Block | 99
  3rd Degree AV block | 147
Sick Node Dysfunction [Number; unit: participants]
  Sick Node Dysfunction | 205
  No Sick Node Dysfunction | 261
Neurocardiogenic Syncope [Number; unit: participants]
  Previous Neurocardiogenic Syncope | 75
  No Previous Neurocardiogenic Syncope | 391

OUTCOME MEASURES:

1. Primary Outcome: Freedom From RA and RV Lead-related Complications
Description: Safety of the Accent MRI™ system with the Tendril MRI™ lead will be evaluated in terms of freedom from Right Atrial (RA) and Right Ventricular (RV) lead-related complications for the acute (implant to 2 month visit) and chronic (2 month visit through the 12 month visit) timeframes.
Time Frame: up to 12 months post-implant
Population: A total of 464 patients were implanted. 463 patients (99.78%) were implanted with Accent MRI™ systems with the Tendril MRI™ leads while the remaining 1 patient (0.22%) was implanted with a device that was not an Accent MRI™ system. This patient was excluded from all primary endpoint analyses.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Accent MRI System
Number analyzed (Participants) | 463
percentage of participants
  Acute Timeframe (Implant to 2 Months) | 97.19 [94.94 to 98.63]
  Chronic Timeframe (>2 Months to 12 Months) | 99.14 [97.58 to 99.81]

ADVERSE EVENTS:
Time Frame: Data collection on adverse events were collected from Enrollment until 12M follow up, i.e. 1 year.
Arm/Group | Accent MRI System
Serious Adverse Events (participants affected / at risk) | 174/466
Other Adverse Events (participants affected / at risk) | 78/466
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accent MRI System (N=466)
Arrhythmia (Cardiac disorders) | 25 (25)
Cardiac/Venous Perforation (Vascular disorders) | 2 (2)
Device migration (Surgical and medical procedures) | 1 (1)
Exacerbation of Diabetes (Endocrine disorders) | 2 (2)
Exacerbation of heart failure (Cardiac disorders) | 15 (15)
Helix issue (Surgical and medical procedures) | 1 (1)
hematoma/bleeding (Injury, poisoning and procedural complications) | 5 (5)
Impedance out of range (Surgical and medical procedures) | 1 (1)
infection (Infections and infestations) | 20 (20)
lead dislodgement or migration (Surgical and medical procedures) | 12 (12)
Muskuloskeletal event (Musculoskeletal and connective tissue disorders) | 10 (10)
Lead replacement (Surgical and medical procedures) | 1 (1)
neoplastic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
neurological event (Nervous system disorders) | 16 (16)
other various (Investigations) | 16 (16)
Other Cardiac/cardiovascular (Cardiac disorders) | 26 (26)
Other lead related (Surgical and medical procedures) | 1 (1)
Pneumothorax/hemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary events (Respiratory, thoracic and mediastinal disorders) | 9 (9)
renal event (Renal and urinary disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accent MRI System (N=466)
arrhythmia (Cardiac disorders) | 27 (27)
Decreased right ventricular sensing (Investigations) | 1 (1)
device programming (Investigations) | 2 (2)
exacerbation of heart failure (Cardiac disorders) | 4 (4)
hematoma/bleeding (Injury, poisoning and procedural complications) | 4 (4)
impedance out of range (Investigations) | 2 (2)
infection (Infections and infestations) | 2 (2)
lead noise (Investigations) | 3 (3)
musculoskeletal event (Musculoskeletal and connective tissue disorders) | 3 (3)
neurological event (Nervous system disorders) | 3 (3)
other various (Investigations) | 13 (13)
other cardio/cardiovascular (Cardiac disorders) | 9 (9)
Other lead related (Investigations) | 1 (1)
Pacemaker software issue (Investigations) | 1 (1)
pulmonary event (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less